CLINICAL TRIAL: NCT01389804
Title: Parents of Pediatric Solid Organ Transplant Recipients: Transition to Home and Chronic Illness Care
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Stacee Lerret, Assistant Professor, Medical College of Wisconsin
Other Study IDs: CHW10/115,GC 1127
Record Dates: First submitted 2010-09-03; First posted 2011-07-08 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Transplant
Keywords: transplant, pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Solid Organ Transplant: Parents of pediatric solid organ transplant recipients

SUMMARY:
The overall long term objective of this research is to improve health care utilization and quality of life of pediatric solid organ transplant recipients and family. Understanding the process of transition to a chronic medical condition during the acute (3 weeks after transplant) and long term (3 and 6 months) will significantly guide the development of clinical interventions aimed at maximizing adherence and family psychosocial adjustment.

DETAILED DESCRIPTION:
Parents of children that have received a heart, kidney, liver or lung transplant will be invited to participate in this protocol.

Involvement in this study entails completion of questionnaires at 4 separate time points. Parents will first complete questionnaires regarding discharge teaching, care coordination and readiness for hospital discharge on the day of discharge from the hospital. Parents will subsequently complete questionnaires at 3 weeks, 3 months and 6 months after discharge. The post discharge questionnaires assess coping, family management, adherence and utilization of healthcare resources.

Currently, no research has been conducted related to readiness for hospital discharge of a parent as the primary caregiver for a child with solid organ transplant or the sequential relationships between hospitalization care and the trajectory of post-discharge outcomes. This research will fill the gap in knowledge needed for care of solid organ transplant children and parents.

The ability to identify factors in the first year after transplant that are predictive of decreased coping and non-adherence affords an opportunity to develop nursing and health interventions that have significant implications for care decisions, as well as disease activity and health care costs.

ELIGIBILITY:
Inclusion Criteria:

1. the parent's child has undergone a heart, kidney, liver, lung or multivisceral transplant and is being discharged home from the hospital
2. the parent is English speaking (tools being used have been validated for English participants only)
3. the parent is 18 years of age or older

Exclusion Criteria:

1. presence of significant communication or cognitive impairment on the part of the parent that would preclude completion of questionnaires based on self-report
2. the child has already experienced the discharge to home transition after a previous transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of pediatric solid organ transplant recipients (heart, kidney, liver or lung)
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Determine if discharge preparation has an effect on parent readiness for hospital discharge and if readiness for hospital discharge effects post-discharge outcomes following hospital discharge in parents of solid organ transplant recipients | 2 years
  Determine if discharge preparation (discharge teaching and care coordination) for parents of solid organ transplant children has an effect on:
  (1) short term discharge transition outcomes and transition to home-based care (measured at 3 weeks post-discharge) and,(2) longer term chronic care outcomes at 3 and 6 months post-discharge.

SECONDARY OUTCOMES:
Post transplant outcomes | 2 years
  Determine outcomes (parent coping, adherence, family management, and utilization of healthcare services) and the relationship between these outcomes, throughout the transition to chronic care management for families of solid organ transplant recipients at 3 weeks, 3 months and 6 months post-discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Stacee Lerret, PhD(c), RN, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin
Locations (5):
- United States (5):
  - Children's Memorial Hospital, Chicago, Illinois
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital and Medical Center of Nebraska, Omaha, Nebraska
  - Levine Children's Hospital, Charlotte, North Carolina
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin